CLINICAL TRIAL: NCT01475435
Title: Oxidative Stress Markers Evaluation Before and After Periodontal Treatment of Diabetics Type 2 Patients With Generalized Chronic Periodontitis and Healthy Periodontium
Brief Title: Oxidative Stress Markers Evaluation Before and After Periodontal Treatment of Diabetics Type 2 Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Antonio Pugliesi Alves de Lima, Associate professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DMSAL2712
Record Dates: First submitted 2011-08-22; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- chronic periodontitis (Active Comparator): Saliva and GCF samples will be evaluated before and after treatment from patients treated of chronic periodontitis.
  Interventions: Procedure: non- surgical periodontal treatment
- periodontally healthy individuals (Placebo Comparator): Saliva and GCF samples will be evaluated from periodontally healthy individuals at baseline.
  Interventions: Procedure: Prophylaxis
- chronic periodontitis with diabetes type 2 (Active Comparator): Saliva and GCF samples will be evaluated before and after treatment from patients with diabetes type 2 treated of chronic periodontitis
  Interventions: Procedure: non- surgical periodontal treatment
- periodontally healthy individuals with diabetes type 2 (Placebo Comparator): Saliva and GCF samples will be evaluated from periodontally healthy individuals with diabetes type 2 at baseline
  Interventions: Procedure: Prophylaxis

INTERVENTIONS:
Procedure: non- surgical periodontal treatment — scaling and root planning
  Arms: chronic periodontitis; chronic periodontitis with diabetes type 2
Procedure: Prophylaxis — Periodontally healthy patients will receive oral hygiene instructions and prophylaxis.
  Arms: periodontally healthy individuals; periodontally healthy individuals with diabetes type 2

SUMMARY:
Abstract Diabetes mellitus and periodontal diseases are both chronic inflammatory disorders that have a major impact on the health and well being of millions of individuals worldwide. Periodontal diseases are among the most common diseases in humans, therefore, if the presence of periodontal diseases plays any role in overall systemic health, the public health impact may be substantial. An important factor that can be involved in the progression of the periodontal disease is the production of Reactive Oxygen Species (ROS). The imbalance between oxidative stress induced by ROS and the concentrations (or activity) of the antioxidant may result in tissue damage. The ROS induce the activity of lipid peroxidation-Tbars, myeloperoxidase (MPO), peroxidase and arginase, whose mechanisms reflect the severity of the periodontal disease and it may offer the basis for a patient specific diagnostic test for periodontitis and could have therapeutic significance. The aim of this study is to investigate quantitatively the levels of oxidative stress markers (Myeloperoxidase, Peroxidase, Lipid Peroxidation and Arginase) in saliva and in gingival crevicular fluid (GCF) of diabetes type 2 subjects with generalized chronic periodontitis and periodontally healthy individuals, and systematically healthy individuals with generalized chronic periodontitis and periodontally healthy individuals, before and after periodontal treatment. Unstimulated whole saliva will be collected for 5 min as well as GCF of 25 diabetes type 2 with generalized chronic periodontitis, 25 diabetes type 2 periodontally healthy individuals as controls, 25 systematically healthy individuals with generalized chronic periodontitis and 25 periodontally healthy individuals before and after treatment. The following clinical parameters will be evaluated: probing pocket depth, probing attachment level, plaque index and the gingival index. The activity of stress markers in saliva and GFC will be analyzed by spectrophotometry. Adequate statistical analysis will be carried out with a p-value set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes and chronic periodontitis(more than 30% of the sites involved, AAP, 1999)
* Patients with type 2 diabetes and periodontally healthy (AAP, 1999)
* Patients systemically healthy with chronic periodontitis (more than 30% of the sites involved)
* Patients systemically and periodontally healthy
* Patients with at least 15 natural teeth (excluding 3rd molars).
* At least 30% of sites with probing pocket depth (PD)> 5 mm and a maximum of 60% sites with PS <7 mm
* Clinical attachment level (CAL)> 4 mm
* Visible plaque and bleeding on probing (BOP)
* Patients with type 2 diabetes have to bear the disease for at least five years and have to show a blood percentage of glycated hemoglobin between 6.5% to 8% (UKPDS 1998) at baseline

Exclusion Criteria

* Individuals with periodontal pockets deeper than 7 mm
* Patients with any other systemic disease (except diabetes type 2)
* Patients who have used medications such as anticoagulants, contraceptives or antidepressants in the past 6 months
* Patients who have used antibiotic and anti-inflammatory drugs in the last 3 months before the of the study
* Smoking
* Pregnancy
* Patients who have received periodontal treatment in the last six months before the start of this study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate level change of oxidative stress biomarkers in crevicular gingival fluid and whole saliva on diabetes type 2 individuals | baseline and 4 weeks after periodontal treatment
  The participants will be followed for an expected average of 4 weeks after periodontal treatment. The samples of saliva and crevicular gingival fluid will be evaluated at baseline and four weeks after periodontal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz A Lima, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil